CLINICAL TRIAL: NCT03627169
Title: PSG Validation of MATRx Plus AHI
Status: Completed | Type: Observational
Sponsor: Zephyr Sleep Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: ZCP201704
Record Dates: First submitted 2018-08-02; First posted 2018-08-13 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MATRx plus/PSG group: Healthy individuals, individuals suspected of having OSA, and individuals with a previous diagnosis of OSA will spend a single night in a sleep laboratory and undergo a standard polysomnogram simultaneously with a Level III sleep study using the MATRx plus device. There is no interventional aspect to the study.
  Interventions: Device: MATRx plus

INTERVENTIONS:
Device: MATRx plus — The MATRx plus device will be used in its capacity as a Level III home sleep apnea test (HSAT). Note: MATRx plus is approved for use in Canada; therefore, the study does not involve any investigational devices.

SUMMARY:
Obstructive sleep apnea (OSA) is a common disease that carries significant risks for cardiovascular disease, mortality, and economic costs. Almost thirty years ago, initial population studies found the prevalence of OSA to be five to nine percent of the adult population. Excess body weight is a risk factor for the development of OSA, and the recent rise in prevalence of obesity has led to revised estimates of OSA prevalence, now at seventeen per cent of the adult population. OSA is poorly recognized clinically; 85% of apneics remain undiagnosed and untreated.

Currently, the diagnosis of OSA commonly relies on an overnight, in-hospital polysomnogram (PSG). Due to the extensive attachments to the body surface required in a PSG, it has developed a negative impression. Any effective solution to the public health challenges posed by sleep apnea will have to consider the need for less cumbersome and off-putting methods.

Zephyr Sleep Technologies has developed a device that has been approved for use in Canada. The MATRx plus device functions as both a Level III sleep recorder (records respiratory airflow, respiratory effort, pulse rate, and arterial oxygen saturation) as well as a home-based system to select patients for oral appliance therapy. The American Academy of Sleep Medicine (AASM) recommends the use of apnea-hypopnea index (AHI) for the diagnosis and categorization of OSA severity. The Level III function of the MATRx plus device is approved for use in Canada with two autoscoring methods: oxygen desaturation index, ODI and apnea-hypopnea index, AHI, but requires further validation of AHI for clearance by the US Food and Drug Administration (FDA).

The proposed research will validate the AHI autoscoring function of the MATRs plus Level III home sleep recorder by comparing it to data recorded in a PSG, which is considered to be the gold standard for sleep testing. Though the effectiveness of the AHI autoscoring algorithm has been previously established, it has not been validated against PSG data. Additionally, other parameters such as snoring will be examined in order to develop scoring algorithms for other facets of sleep disordered breathing.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disease that carries significant risks for cardiovascular disease, mortality, and economic costs. Almost thirty years ago, initial population studies found the prevalence of OSA to be five to nine percent of the adult population. Excess body weight is a risk factor for the development of OSA, and the recent rise in prevalence of obesity has led to revised estimates of OSA prevalence, now at seventeen per cent of the adult population. OSA is poorly recognized clinically; 85% of apneics remain undiagnosed and untreated.

OSA derives fundamentally from structural abnormalities of the pharynx that cause pharyngeal narrowing or closure during sleep and produce recurrent apneas and hypopneas. During wakefulness, compensatory neuromuscular reflexes protect the pharynx from collapse. These reflexes are lost during sleep, leaving the collapsible human pharynx susceptible to narrowing or closure. Owing largely to its association with excess body weight, OSA has arguably become the most prevalent chronic non-communicable disease in industrialized societies, assuming that obesity is not classified a disease. In addition to impairing quality of life, OSA conveys an increased risk of cardiovascular disease and vehicular accidents. The majority of apneics remain undiagnosed and untreated. Thus, OSA has the hallmarks of a major public health problem, affecting all age groups and increasing in epidemic proportions. Unfortunately, current medical practices seem ill-suited to dealing with the challenges posed by OSA.

Perhaps the most unsettling aspect of present medical practices relates to the cumbersome, uninviting, and expensive methods currently used to diagnose the disease. Common clinical experience indicates that individuals often resist undergoing the standard diagnostic test, an overnight in-hospital polysomnogram (PSG), because of the extensive attachments to the body surface. In other words, as public awareness of sleep apnea has increased so also has the negative impression of current testing. Any effective solution to the public health challenges posed by sleep apnea will have to consider the need for less cumbersome and off-putting clinical methods.

Zephyr Sleep Technologies has developed a device that has been approved for use in Canada. The device, MATRx plus, functions as both a Level III sleep recorder (records respiratory airflow, respiratory effort, pulse rate, and arterial oxygen saturation) as well as a home-based system to select patients for oral appliance therapy. The American Academy of Sleep Medicine (AASM) recommends the use of apnea-hypopnea index (AHI) for the diagnosis and categorization of OSA severity. The Level III function of the MATRx plus device is approved for use in Canada with two autoscoring methods: oxygen desaturation index, ODI and apnea-hypopnea index, AHI, but requires further validation of AHI for clearance by the US Food and Drug Administration (FDA).

The proposed research will validate the AHI autoscoring function of the MATRs plus Level III home sleep recorder by comparing it to data recorded in a PSG, which is considered to be the gold standard for sleep testing. Though the effectiveness of the AHI autoscoring algorithm has been previously established, it has not been validated against PSG data. Additionally, other parameters such as snoring will be examined in order to develop scoring algorithms for other facets of sleep disordered breathing.

Once the participant arrives at the PSG laboratory, the clinical coordinator will obtain written informed consent, review inclusion and exclusion criteria, and enroll eligible participants into the study. The clinical coordinator will give the participant a brief overview on use of the MATRx plus Level III sleep recorder, then return to the control room to watch the participant set up the device via video. The participant will be made aware of the video recorded during set up the MATRx plus device. The device set up consists of: dual nares nasal cannula for airflow, respiratory effort belt, pulse oximeter, snoring (recorded via airflow frequency on the nasal cannula and via sound on the tablet), body position from an accelerometer built into the body-worn recorder. The sleep technician will then set the participant up with a standard PSG montage, consisting of: electroencephalogram (EEG), electrooculogram (EOG), electromyogram (EMG), pulse oximeter, nasal cannula, two respiratory effort belts, snoring, and body position (recorded via body-mounted accelerometer). Once the participant has both the MATRx plus and the PSG montage set up, the study will commence, and the participant will be monitored by video from the PSG control room, as is standard practice in a PSG. The sleep technician will intervene as necessary to ensure adequate signals are collected by the PSG equipment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21 and 80 years
* Ability to understand and provide informed consent
* Ability and willingness to meet the required schedule

Exclusion Criteria:

* Inability to breathe comfortably through the nose
* Symptomatic, non-respiratory sleep disorder, e.g., restless leg syndrome, chronic insomnia
* Heart failure
* Cerebral vascular incident within the last 12 months
* Use of pacemaker or other life-supporting device

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals, individuals who suspect they may have OSA, and individuals who have previously been diagnosed with or treated for OSA will be recruited for the trial. Only participants who meet all eligibility criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Apnea and hypopnea events | 1 night
  The number of apnea and hypopnea events collected from each the MATRx plus device and PSG will be recorded in order to determine the sensitivity/specificity of the MATRx plus device.

SECONDARY OUTCOMES:
Snoring events | 1 night
  The number of snoring events

CONTACTS AND LOCATIONS:
Locations (1):
- Zephyr Sleep Technologies, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers.

REFERENCES:
- [Derived] Topor ZL, Remmers JE, Grosse J, Mosca EV, Jahromi SAZ, Zhu Y, Bruehlmann S. Validation of a new unattended sleep apnea monitor using two methods for the identification of hypopneas. J Clin Sleep Med. 2020 May 15;16(5):695-703. doi: 10.5664/jcsm.8324. Epub 2020 Feb 6. PMID 32024586